CLINICAL TRIAL: NCT01995214
Title: Comparison of Sevoflurane and Propofol Anesthesia on Postoperative Delirium in Geriatric Patients
Brief Title: Sevoflurane and Propofol Anesthesia on Postoperative Delirium
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Associate Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TJMZK20130602
Record Dates: First submitted 2013-11-13; First posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: General Anesthesia; Geriatric Patient
Keywords: Postoperative delirium; Geriatric; General anesthesia; Propofol; Sevoflurane
MeSH Terms: conditions — Emergence Delirium | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- P (Experimental): Anesthesia maintenance with propofol+remifentanil
  Interventions: Drug: Propofol
- S (Experimental): Anesthesia maintenance with sevoflurane+remifentanil
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Anesthesia maintenance with propofol+remifentanil guided by Narcotrend index monitoring.
  Arms: P
Drug: Sevoflurane — Anesthesia maintenance with sevoflurane+remifentanil guided by Narcrotrend index monitoring.
  Arms: S

SUMMARY:
Delirium is defined as an acute onset and fluctuating course of mental status change with inattention and an altered level of consciousness. Delirium in the postoperative period can be divided into emergence delirium and postoperative delirium, based on the time of onset (Silverstein et al., 2007).Postanaesthesia delirium is a frequent and potentially serious problem affecting the safety of patients and medical personnel. Clinical studies demonstrated that postoperative delirium is associated with worse outcomes such as prolonged hospital stay, postdischarge institutionalization, and increased mortality (Ely et al., 2004a; Thomason et al., 2005; Robinson et al., 2009). Multiple factors may contribute to the development of postoperative delirium, including patient's medical condition, administration of anesthetics or analgesics and degree of operative stress (Yildizeli et al., 2005; Robinson & Eiseman, 2008; Deiner & Silverstein, 2009). Sevoflurane anesthesia have been reported to be associated with more emergence delirium in pediatric patients, when compared with propofol anesthesia. It is not clear if propofol anesthesia will benefit the geriatric patients on postoperative delirium, when compared with sevoflurane anesthesia. We hypothesize that propofol anesthesia will reduce the rate of postoperative delirium by 50% when compared with sevoflurane anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Status classification (ASA_PS) class I-III
* Aged 60 years or above
* Elective major surgery under general anesthesia

Exclusion Criteria:

* ASA_PS>=IV
* Aged under 60 yr old
* Body mass index (BMI) >30
* Neurologic disease
* Cardiac surgery and neurologic surgery
* Anticonvulsant drugs
* Chronic analgesics intake
* Participating in the investigation of another study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium | at 24 postoperative hours
  Postoperative delirium was determined by Confusion Assessment Method (CAM) at 24 postoperative hours

SECONDARY OUTCOMES:
Length of postanesthesia care unit (PACU) stay | up to 2 hours after PACU admitting
  Length of PACU stay (min)
Hemodynamic parameters | 5min, 10min, 20min, 30min after induction, 5min, 10min, 20min, 30min after skin incision, 5min, 10min, 20min, 30min before incision closure
  Hart frequency, systolic blood pressure, diastolic blood pressure
Incidence of postoperative nausea and vomiting | 24 postoperative hours
  Incidence of postoperative nausea and vomiting
Quality of recovery determined by quality of recovery (QOR-40; maximum score 200) score | 1,2,3,7 postoperative days
  Quality of recovery determined by QOR-40
Postoperative delirium | 2st, 3st, 7st postoperative days
  Postoperative delirium was determined by CAM every day at 2st, 3st, 7st postoperative days
Postoperative Stroke | 1st, 2st, 3st, 7st postoperative days
  Postoperative Stroke will be determined by National Institutes of Health Stroke Scale (NIHSS)

CONTACTS AND LOCATIONS:
Overall Officials: Yuke Tian, MD., PhD., Study Chair — Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China